CLINICAL TRIAL: NCT04478669
Title: Optimal Imaging Methods to Reduce Repeat Surgery in Invasive Breast Cancer
Brief Title: Digital Breast Tomosynthesis (DBT) to Improve Assessment of Resection Margins in Invasive Breast Cancer
Acronym: DBT
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Irina Palimaru Manhoobi, MD, PhD student, radiologist, Aarhus University Hospital
Other Study IDs: 1107210020
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Invasive Breast Cancer; Mastectomy, Segmental; Margins of Excision
Keywords: Digital breast tomosynthesis; Diagnostic imaging
MeSH Terms: conditions — Margins of Excision

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The challenge of breast conserving surgery (BCS) is to obtain free resection margins, by removing the invasive tumor and the precursor cells: DCIS (Ductal Carcinoma in Situ). Consequently, 17%-25% of primary invasive breast cancer patients will need a repeat surgery. Repeat breast surgery has been associated with higher surgical risks, poorer cosmetic outcome and increased psychological and economic burden. Finding a precise method to obtain tumor- and DCIS-free resection margins during BCS is therefore strongly needed.

The purpose with this study is to investigate if the need for a re-operation can be reduced by performing Digital Breast Tomosynthesis (DBT) of the resected tumor margins compared to the currently used standard X-ray during BCS.

DETAILED DESCRIPTION:
Background Breast cancer is the most common type of cancer in Denmark with approximately 4700 new cases each year, with an increased incidence during the last decades. Almost 70% of the patients are treated with breast conserving surgery (BCS) and breast irradiation. Unfortunately, 5.9 % of the patients treated with BCS will experience local recurrence after 9 years. The strongest predictor for local recurrence is a positive pathologic resection margin. Therefore it is important intraoperatively to be able to evaluate the margin width of the resected specimen precisely. The challenge during BCS is to remove the primary invasive breast cancer, with negative resection margin, free of invasive tumor and DCIS, Ductal Carcinoma In Situ. Some have concluded that lack of accurate imaging especially of the DCIS is the main reason for positive margins and repeat surgery, as the DCIS often, but not in all cases, contains microcalcifications that can be detected on mammography (x-ray of the breast). Consequently, 17%-25% of the patients will need a second or a third surgery. Repeat surgery has been associated with higher surgical risk, poorer cosmetic outcome, and increased psychological and economic burden for both patients and the society. Finding an optimal imaging method to obtain adequate resection margins close to or during BCS that can reduce the number of repeat surgeries, is therefore strongly needed.

Definition of resection margin status

A safe macroscopic surgical resection margin is, according to the Danish Breast Cancer Group´s (DBCG) guidelines, defined as a margin width ≥ 5mm minimizing the risk of leaving residual tumor. In many institutions in Denmark, a perioperative evaluation of the tumor is performed as a macroscopically assessment by a pathologist. This is a ressource demanding procedure and X-ray of the specimen is used instead. A radiological, positive resection margin is defined as a margin width of 0 mm, that leads to a re-excision during the same surgical procedure, and additional breast tissue is removed at the exact same area of the patient's breast. This procedure aims to avoid the discomfort of a repeat surgery. The perioperative radiological assessment of the resection margins is afterwards confirmed microscopically, where a positive margin at our institution is defined as "tumor on ink", meaning tumor cells in the inked resection margin with 0 mm to the margin. A positive margin will trigger a repeat surgery, either a new BCS or a mastectomy where the whole breast is removed. For DCIS, a margin-width of less than 2 mm is considered positive, and the patient will be offered repeat surgery according to guidelines. A distance from the invasive carcinoma to the resection margin of < 2 mm, but not "on the ink" is surgical considered sufficient and the patient will according to DBCG guidelines, not require a repeat surgery, but will instead be offered additional boost to the subsequent radiotherapy. The result of the final histopathology is, however, not available until 7 workdays after the initial BCS. Guidance of a more optimal perioperative methods to evaluate the resection margins during BCS would, therefore, be highly desirable, and could potentially lead to a decreased rate of repeat surgery and hence save several patients from the discomfort of a second surgical procedure.

Intraoperative imaging methods for margin assessment

Various methods to assess resection margins have been investigated such as frozen section analysis, imprint cytology, macroscopically evaluation and imaging with x-ray, micro-CT scanning or ultrasound of the resected tumor margins. All have, however, their limitations, either because they are time consuming, or simply because they are not accurate enough to predict resection margin status. The imaging modality X-ray has been reported in several studies to have a high specificity, predicting negative margins up to 95%, but unfortunately a low sensitivity of only 21%. That means that the method is particularly good to predict a negative margin. The X-ray is less sensitive when it comes to predict a positive resection margin, with the final histopathology as a reference method. The lower sensitivity is due to the fact, that x-ray has difficulties, when it comes to detect the breast tumor in a very dense normal breast tissue, most common for young women. The X-ray evaluation also has the disadvantage of only delivering a 2D solution to a 3D problem. The other imaging method currently in use is ultrasound that has a high sensitivity of 80% but a low specificity of 59% to predict positive resection margins (Ramos M. et al).

A new method called Micro-CT (micro-Computed Tomography) can provide 3D imaging of the resected tumor and the microcalcifications that helps to asses all margins of the resected tumor. Unfortunately, there is a high interobserver variability reported with this method. Furthermore, it is difficult to differentiate between tumor and normal breast tissue in the resected margins in some of the cases, which makes it impossible for the radiologist to determine if the margins are positive or negative. This may be one of the reasons for, why this method does not perform so well with a sensitivity range of only 38%-56%.

Digital Breast Tomosynthesis (DBT) is a novel method for assessment of resection margins based on X-ray technology. DBT provides images of the resected tumor with a large field of view of the specimen and a high resolution, that allows the radiologist to examine the resected specimen in one millimeter increments both in 2D and 3D, where the extent and the shape of the tumor and the microcalcifications are better defined than on conventional 2D mammography. Only few clinical studies have investigated DBT for evaluation of resection margins with the most recent study with 98 patients included (Park KU. et al). This study reported a high performance of the DBT with a sensitivity to predict positive margins of 93%, and a specificity of 78%, to predict negative margins, with the final histopathology as a reference method.

Objectives

The overall objective of the present study is to investigate if adequate resection margins can be obtained with use of DBT of the resected margins during BCS to reduce the rate of repeat surgery and avoid further unnecessary complications and psychological stress for the patients.

Hypothesis

Does intraoperative DBT improve assessment of the resected margins compared to standard method with X-ray? The final histopathology will be used as a reference method.

1. DBT can contribute to obtain negative resection margins and thereby reduce the need of repeat surgery as compared to X-ray.
2. The performance of DBT predicting resection margin status is more accurate compared to the standard method with X-ray.

Study participants

The study participants will be recruited at the Department of Plastic and Breast Surgery at Aarhus University Hospital after they have been diagnosed with operable invasive breast cancer and scheduled for BCS. The study participants will receive separate information leaflet about this project that respects the applicable regulatory requirements. The page describing the rights of the patient participating in a health research project will also be handed out to the patient by the breast surgeon. The breast surgeon will obtain the informed consent from the patient and mention in the patient's medical record, that the patient has given consent to participate in this project.

Randomization

The study participant will be randomized to either the DBT or the standard method (X-ray) by the breast surgeon in the system REDCap®. REDCap® is a secure web platform that can build and manage online databases and surveys that will also be used for the data management of this project. The randomization will be performed by the breast surgeon during the first consultation with the patient, as soon as the patient has given oral and written consent and is included in each trial.

Handling of the resected breast tumor

The study encompasses tissue being procured as part of the normal diagnostic procedure. The material will, as all tissue collected for diagnostic purposes, be kept in the existing clinical biobank at the Department of Pathology, at Aarhus University Hospital during as well as after the closure of the study. A research biobank will therefore not be established

Safety

There are no side effects and no risk of radiation for the investigators in the DBT-trial, as the resected tumor will be located inside the DBT or in the X-ray that is a closed system, ex-vivo, with no radiation exposure to the technical staff or to the study patients.

Statistics and analysis

A sample size of 123 study participants was calculated as necessary to detect a reduction from 20% in the X-ray-group to 7% in the DBT-group with a statistical power of 80% and a 5% level of significance. The investigators expect a few patients may drop-out for different reasons, and estimated that a total number of 250 patients are enough to be included in the DBT-trial.

The statistical analyses and calculation will be made primarily by the investigator Irina Palimaru Manhoobi (IPM) using STATA® where after the work will be reviewed by a statistician to ensure a high quality of the statistical work.

1. The occurrence of positive resections margins, re-excisions and repeat surgery will be compared between groups using the Fisher exact test.
2. The performance of the tested and the standard method: The sensitivity, specificity, Positive Predictive Value (PPV) and the Negative Predictive Value (NPV) compared to the reference method will be calculated with the McNemar Chi-Square test.

A two-sided p-value of less than 0.05 will be considered statistically significant.

Data management

The study participants will be identified from the Central Personal Register system (CPR) with permission obtained the 1st of April 2020 from the Danish Data Protection Agency (DDPA) / "Region Midtjyllands interne fortegnelse over forskningsprojekter" with case number 1-16-02-141-20. The informed consent from all study participants gives the investigator, sponsor and the representants of the sponsor, the direct access to the below described clinical data from the medical record (EPJ) Electronical Patient Journal, that is important to perform this project. All clinical data will be transferred anonymously to the secure web application for data management in "RedCap" that is administered by Aarhus University. The investigator IPM is responsible for the data management. The study is in according to the guidelines of the Helsinki Declaration II, GCP guidelines and the Danish Legislation regarding clinical trials and legislation regarding personal data.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed women with biopsy-verified invasive breast cancer planned for breast conserving surgery.
* Age > 18 year

Exclusion Criteria:

* Previous surgery for pre-malignant or malignant lesions in the breast
* Planned mastectomy

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited at the Department of Plastic and Breast Surgery at Aarhus University Hospital after they have been diagnosed with operable invasive breast cancer and scheduled for breast conserving surgery.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Positive resection margin(s) in the final histopathology | 7 workdays, time from primary breastconserving surgery to the time where the final histopathology result is available.
  The number of patients with one or more positive resection margins in the final histopathology.
Re-excision-rate during primary breast conserving surgery | One workday, time from primary breastconserving surgery to the time where data of the re-excision of the cavity during same surgery is available in the patient electronical journal
  The number of patients that recieves further excision of the cavity wherefrom the breast tumor is resected, during the initial breast conserving surgery.
Rate of repeat surgery | 3 weeks from primary breastconserving surgery, depending on the final histopathology result.
  The number of patients that recieves a second or a third surgery due to insufficient resection margins during initial primary breast conserving surgery.

SECONDARY OUTCOMES:
Diagnostic performance of the tested method to predict correct resection margins status. | one year from primary breast conserving surgery, when the inclusion of all patients is final and the dataanalysis is ready.
  Sensitivity, specificity, positive and negative predictive value and accuracy of the tested method to predict accurate resection margin status.
Weight of the re-excised breast tumor during initial breast conserving surgery | One work day, The weight will be registered during the day the patient recieves primary breast conserving surgery and will be registered by the surgeon in the patient electronical journal.
  The weight of the re-excised breast tumor during initial breast conserving surgery to see if there is a difference of how much tissue is removed with the tested method DBT and the standard X-ray method.
Type of repeat surgery (both secondary and if any tertiar surgery) | 3 weeks from the primary breastconserving surgery, depending on the final histopathology result and what type of repeat surgery the patient is planned to recieve
  The type of repeat surgery, either breast conserving surgery or mastectomy where the whole breast is removed.

CONTACTS AND LOCATIONS:
Overall Officials: Peer Christiansen, DMSc, Prof., Principal Investigator — Department of Plastic and Breast Surgery, Aarhus University Hospital
Locations (1):
- Department og Plastic- and Breast Surgery, Aarhus, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Amiel CR, Fisher HM, Carver CS, Antoni MH. The importance of stress management among postresection breast cancer patients. Future Oncol. 2016 Dec;12(24):2771-2774. doi: 10.2217/fon-2016-0442. Epub 2016 Oct 19. No abstract available. PMID 27756150
- [Background] DeSnyder SM, Hunt KK, Dong W, Smith BD, Moran MS, Chavez-MacGregor M, Shen Y, Kuerer HM, Lucci A. American Society of Breast Surgeons' Practice Patterns After Publication of the SSO-ASTRO-ASCO DCIS Consensus Guideline on Margins for Breast-Conserving Surgery With Whole-Breast Irradiation. Ann Surg Oncol. 2018 Oct;25(10):2965-2974. doi: 10.1245/s10434-018-6580-9. Epub 2018 Jul 9. PMID 29987598
- [Background] Thill M, Baumann K, Barinoff J. Intraoperative assessment of margins in breast conservative surgery--still in use? J Surg Oncol. 2014 Jul;110(1):15-20. doi: 10.1002/jso.23634. Epub 2014 May 24. PMID 24863286
- [Result] Bodilsen A, Bjerre K, Offersen BV, Vahl P, Amby N, Dixon JM, Ejlertsen B, Overgaard J, Christiansen P. Importance of margin width in breast-conserving treatment of early breast cancer. J Surg Oncol. 2016 May;113(6):609-15. doi: 10.1002/jso.24224. Epub 2016 Mar 16. PMID 26991020
- [Result] Smitt MC, Nowels K, Carlson RW, Jeffrey SS. Predictors of reexcision findings and recurrence after breast conservation. Int J Radiat Oncol Biol Phys. 2003 Nov 15;57(4):979-85. doi: 10.1016/s0360-3016(03)00740-5. PMID 14575828
- [Result] Jeevan R, Cromwell DA, Trivella M, Lawrence G, Kearins O, Pereira J, Sheppard C, Caddy CM, van der Meulen JH. Reoperation rates after breast conserving surgery for breast cancer among women in England: retrospective study of hospital episode statistics. BMJ. 2012 Jul 12;345:e4505. doi: 10.1136/bmj.e4505. PMID 22791786
- [Result] Bodilsen A, Bjerre K, Offersen BV, Vahl P, Ejlertsen B, Overgaard J, Christiansen P. The Influence of Repeat Surgery and Residual Disease on Recurrence After Breast-Conserving Surgery: A Danish Breast Cancer Cooperative Group Study. Ann Surg Oncol. 2015 Dec;22 Suppl 3:S476-85. doi: 10.1245/s10434-015-4707-9. Epub 2015 Jul 16. PMID 26178760
- [Result] McCahill LE, Single RM, Aiello Bowles EJ, Feigelson HS, James TA, Barney T, Engel JM, Onitilo AA. Variability in reexcision following breast conservation surgery. JAMA. 2012 Feb 1;307(5):467-75. doi: 10.1001/jama.2012.43. PMID 22298678
- [Result] Hisada T, Sawaki M, Ishiguro J, Adachi Y, Kotani H, Yoshimura A, Hattori M, Yatabe Y, Iwata H. Impact of intraoperative specimen mammography on margins in breast-conserving surgery. Mol Clin Oncol. 2016 Sep;5(3):269-272. doi: 10.3892/mco.2016.948. Epub 2016 Jul 4. PMID 27588192
- [Result] Ramos M, Diaz JC, Ramos T, Ruano R, Aparicio M, Sancho M, Gonzalez-Orus JM. Ultrasound-guided excision combined with intraoperative assessment of gross macroscopic margins decreases the rate of reoperations for non-palpable invasive breast cancer. Breast. 2013 Aug;22(4):520-4. doi: 10.1016/j.breast.2012.10.006. Epub 2012 Oct 27. PMID 23110817
- [Result] McClatchy DM 3rd, Zuurbier RA, Wells WA, Paulsen KD, Pogue BW. Micro-computed tomography enables rapid surgical margin assessment during breast conserving surgery (BCS): correlation of whole BCS micro-CT readings to final histopathology. Breast Cancer Res Treat. 2018 Dec;172(3):587-595. doi: 10.1007/s10549-018-4951-3. Epub 2018 Sep 17. PMID 30225621
- [Result] Park KU, Kuerer HM, Rauch GM, Leung JWT, Sahin AA, Wei W, Li Y, Black DM. Digital Breast Tomosynthesis for Intraoperative Margin Assessment during Breast-Conserving Surgery. Ann Surg Oncol. 2019 Jun;26(6):1720-1728. doi: 10.1245/s10434-019-07226-w. Epub 2019 Mar 14. PMID 30877499